CLINICAL TRIAL: NCT07110246
Title: A Phase 2 De-escalation Study of Dabrafenib and Trametinib for Patients With BRAF V600 Mutant Low-Grade Gliomas
Brief Title: Dabrafenib and Trametinib for BRAF V600 Mutant Low-Grade Gliomas
Acronym: PNOC037
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25081; NCI-2025-04985 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: BRAF V600 Mutation; Low-grade Glioma; Low Grade Glioma of Brain; Recurrent Low Grade Glioma
MeSH Terms: interventions — dabrafenib; trametinib; Magnetic Resonance Spectroscopy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Arm A (Newly diagnosed, Dabrafenib, Trametinib followed by treatment stop) (Experimental): Participants with newly diagnosed BRAF V600 mutant LGGs receive dabrafenib PO twice per day (BID) and trametinib PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for a minimum of 12 cycles and continues until confirmed best response or for up to a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity. Participants then stop treatment with dabrafenib and trametinib. Participants also undergo ECHO, MRI, and blood sample collection throughout the study and may optionally undergo lumbar puncture for collection of CSF.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Specimen Collection; Procedure: Optional Lumbar puncture
- Cohort 1: Arm B (Newly diagnosed, Dabrafenib, Trametinib followed by weaning) (Experimental): Participants with newly diagnosed BRAF V600 mutant LGGs receive dabrafenib PO twice per day (BID) and trametinib PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for a minimum of 12 cycles and continues until confirmed best response or for up to a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity. Participants then receive dabrafenib PO BID and trametinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Participants also undergo ECHO, MRI, and blood sample collection throughout the study and may optionally undergo lumbar puncture for collection of CSF.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Specimen Collection; Procedure: Optional Lumbar puncture
- Cohort 2: Arm A (Recurrent LGG, Dabrafenib, Trametinib followed by treatment stop) (Experimental): Participants with recurrent/progressive BRAF V600 mutant LGGs receive dabrafenib PO twice per day (BID) and trametinib PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for a minimum of 12 cycles and continues until confirmed best response or for up to a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity. Participants then stop treatment with dabrafenib and trametinib. Participants also undergo ECHO, MRI, and blood sample collection throughout the study and may optionally undergo lumbar puncture for collection of CSF.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Specimen Collection; Procedure: Optional Lumbar puncture
- Cohort 2: Arm B (Recurrent LGG, Dabrafenib, Trametinib followed by weaning) (Experimental): Participants with recurrent/progressive BRAF V600 mutant LGGs receive dabrafenib PO twice per day (BID) and trametinib PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for a minimum of 12 cycles and continues until confirmed best response or for up to a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity. Participants then receive dabrafenib PO BID and trametinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Participants also undergo ECHO, MRI, and blood sample collection throughout the study and may optionally undergo lumbar puncture for collection of CSF.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Specimen Collection; Procedure: Optional Lumbar puncture

INTERVENTIONS:
Drug: Dabrafenib — Given orally (PO)
  Other Names: Dabrafenib Mesylate; GSK2118436B; Tafinlar; GSK2118436 Methane Sulfonate Salt
Drug: Trametinib — Given PO
  Other Names: Trametinib Dimethyl Sulfoxide; Mekinist; Meqsel; Spexotras; 1187431-43-1
Procedure: Magnetic Resonance Imaging (MRI) — Undergo imaging by MRI
  Other Names: MRI; MR Imaging
Procedure: Specimen Collection — Under collection of blood and optional CSF samples
  Other Names: Biological Sample Collection
Procedure: Optional Lumbar puncture — Undergo optional lumbar puncture
  Other Names: Optional Spinal tap

SUMMARY:
This phase II trial studies how well de-escalating the drugs dabrafenib and trametinib works in treating patients with low-grade gliomas that have a BRAF V600 gene mutation. Dabrafenib and trametinib are in a class of medications called kinase inhibitors. They work by blocking the action of abnormal proteins that signals tumor cells to multiply. This helps stop the spread of tumor cells. This trial may help doctors determine the best dosing strategy for patients who have received dabrafenib and trametinib for 12-24 months: Either stopping dabrafenib and trametinib completely or slowly reducing the dose for an additional 6 months.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if there is a difference in rate of rebound and/or clinical progression necessitating the reinstitution of treatment at 4 months after stopping or weaning therapy with dabrafenib mesylate (dabrafenib) and trametinib dimethyl sulfoxide (trametinib) in participants with newly diagnosed or recurrent/progressive LGGs with BRAF V600 mutation.

EXPLORATORY OBJECTIVES:

I. To describe the toxicity in participants in different phases of drug administration:

Ia. Standard dosing schedule of dabrafenib and trametinib.

Ib. Abruptly stopping dabrafenib and trametinib.

Ic. Weaning dabrafenib and trametinib.

II. To assess the time to rebound and/or radiologic or clinical progression for participants who abruptly stop dabrafenib and trametinib versus participants who wean dabrafenib and trametinib.

III. To determine the durability of response, defined as time to progression, for patients treated until confirmed best response or for a maximum of 24 months.

IV. To monitor response/toxicity by profiling cell-free deoxyribonucleic acid (DNA) (cfDNA) whole genomes in longitudinal blood and cerebrospinal fluid (CSF) specimens.

V. To correlate response/toxicity based on pharmacogenomics.

VI. To explore response-predictive features in tumor cellular composition and tissue architecture through multi-dimensional data integration (single nucleus multiomics, spatial tumor tissue profiling, digital pathology).

VII. To assess radiogenomic prediction models.

VIII. To assess machine learning imaging models accuracy in evaluating response and compare to standard Response Assessment in Neuro-Oncology Low Grade Glioma (RANO-LGG) and Response Assessment in Pediatric Neuro-Oncology (RAPNO)-LGG criteria.

IX. To describe the microbiome profile in participants receiving dabrafenib and trametinib.

X. To characterize cutaneous toxicities across participants with different skin colors taking a weaning regimen of dabrafenib and trametinib compared to participants taking standard dose dabrafenib and trametinib.

OUTLINE:

Participants receive dabrafenib and trametinib each cycle for a minimum of 12 cycles and up to a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity. Participants are then randomized to 1 of 2 arms.

ARM A: Participants stop treatment with dabrafenib and trametinib.

ARM B: Participants receive dabrafenib PO BID and trametinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed LGG World Health Organization (WHO) Grade I or II with BRAF V600 mutation confirmed by immunohistochemistry or sequencing
* Participants must have measurable tumor.

  * For participants with measurable disease, this will be defined as lesions that can be accurately measured in two dimensions (longest diameter to be recorded) with a minimum size of no less than double the slice thickness. Previously irradiated lesions are considered non-measurable except in cases of documented progression of the lesion since the completion of radiation therapy. Participants without measurable disease may be considered for enrollment and followed for survival and progression purposes but will not be included as part of a measurable disease cohort.
* Cohort 1:

  * Participants must have no prior therapy, except for surgical intervention (i.e. biopsy or resection)
  * Participants may currently be taking dabrafenib and trametinib as frontline therapy, with a maximum duration of 21 months and participants must not yet have met criteria for confirmed best response as defined in this protocol. For participants entering the trial currently taking dabrafenib and trametinib, they must be taking a dose that is within 20% of the standard dosing for both drugs based on age and weight. Participants who are already on dabrafenib and trametinib when enrolling on trial and whose dosing deviates more than 20% from the protocol nomogram need to be discussed with the study chairs. Eligibility for these participants will be based on ability to wean within the parameters of the protocol
* Cohort 2:

  * Participants must have a history of recurrent or progressive disease following prior therapy (e.g., carboplatin and vincristine, vinblastine, bevacizumab, mitogen-activated extracellular signal-regulated kinase (MEK) inhibitor, radiation therapy etc). Participants who previously completed a course of therapy with dabrafenib and trametinib, who did not progress on this therapy, and who are beyond 6 months from completion of therapy are eligible for retreatment.

  ** Participants may currently be taking dabrafenib and trametinib as therapy for disease recurrence, for a maximum duration of 21 months and participants must not yet have met criteria for confirmed best response as defined in this protocol. For participants entering the trial currently taking dabrafenib and trametinib, they must be taking dose that is within 20% of the standard dosing for both drugs based on age and weight. Participants who are already on dabrafenib and trametinib when enrolling on trial and whose dosing deviates more than 20% from the protocol nomogram need to be discussed with the study chairs. Eligibility for these participants will be based on ability to wean within the parameters of the protocol
* Participants must have received their last dose of chemotherapy 3 weeks prior to enrollment (6 weeks for nitrosoureas) and recovered from acute adverse events due to agents administered
* Participants must be at least 7 days since the completion of therapy with a biologic or small molecule agent except dabrafenib and trametinib. For any agent with known adverse events that can occur beyond 7 days after administration, the period prior to enrollment must be beyond the time during which adverse events are known to occur. Such participants must be discussed with study chairs
* Radiation:

  * No prior radiation is allowed for participants in Cohort 1
  * Participants in Cohort 2 must have:

    * Had their last fraction of local irradiation to primary tumor ≥ 12 weeks prior to registration
    * Had their last fraction of craniospinal irradiation ≥ 12 weeks prior to registration
    * At least 14 days after local palliative radiation (small-port)
* Age: ≥ 12 months and < 25 years old
* Performance Score: Karnofsky ≥ 50 for participants > 16 years of age and Lansky ≥ 50 for participants ≤ 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* A serum creatinine ≤ 1.5 upper limit of normal (ULN) based on age and gender
* Total bilirubin ≤ 1.5 x ULN for age; in presence of Gilbert's syndrome, total bilirubin ≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN
* Alanine aminotransferase (ALT) ≤ 3 x ULN
* Aspartate aminotransferase (AST) ≤ 3 x ULN
* Participants with seizure disorder may be enrolled if well controlled
* Left ventricular ejection fraction (LVEF) greater than or equal to institutional lower limit of normal (LLN) by echocardiogram (ECHO) (while not receiving medications for cardiac function)
* Correct QT (QTc) interval < 480 msecs
* Patient must agree to adequate contraception. (The effects of dabrafenib and trametinib on the developing human fetus are unknown. For this reason and because agents as well as other therapeutic agents used on this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method birth control, or abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of the study medication administration. Should a women become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately)
* A legal parent/guardian or patient must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate
* Participants must enroll on Pediatric Neuro-Oncology Consortium (PNOC) comprehensive follow up protocol (PNOC COMP) if PNOC COMP is open to accrual at the enrolling institution
* Pathology reports, next generation sequencing reports, or both, confirming BRAF V600E mutation status must be submitted at the time of enrollment

Exclusion Criteria:

* Participant's tumor has any of the following additional previously known or expected activating molecular alterations:

  * Isocitrate dehydrogenase 1 and 2 (IDH1 and IDH2) mutation
  * Histone H3 mutation (p.K28M, p.G35R, p.G35V)
  * Neurofibromatosis Type 1 (NF-1) loss of function alteration
* Participants who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dabrafenib and trametinib
* Medications that are affected by the induction of CYP3A4 and CYP2C9 should be avoided or used cautiously. Dabrafenib has been shown to induce CYP3A4 and CYP2C9. In addition, dabrafenib is an in vitro inducer of CYP2B6, CYP2C8, CYP2C19, Uridine 5'-diphospho (UDP)-glucuronosyltransferase. Co-administration of dabrafenib and medications which are affected by the induction of these enzymes (including warfarin) and transporters may result in loss of efficacy. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the participant and/or legal parent or guardian will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection
* Women of childbearing potential must not be pregnant or breast-feeding
* Human immunodeficiency virus (HIV) positive participants will be ineligible if HIV therapy regimen has not been stable for at least 4 weeks or there is intent to change the regimen within 8 weeks following enrollment, or if they are severely immunocompromised

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Rebound rate (RR) | Up to a maximum of 34 months
  The Rebound rate is defined as increase in tumor size by 25% or more by Response Assessment in Pediatric Neuro-Oncology-Low Grade Glioma (RAPNO-LGG) criteria and/or clinical progression necessitating the re-institution of therapy occurring within 4 months off therapy for participants with BRAF V600 mutant LGG after abruptly stopping or weaning off dabrafenib and trametinib. RR will be reported by cohort and arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PHD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - John Hopkins Medical Center, Baltimore, Maryland
  - St. Louis Children's Hospital Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be provided to study collaborators during the course of the study
Supporting Information: Study Protocol, SAP, ICF